CLINICAL TRIAL: NCT02748733
Title: Randomized Cross-over Comparison of Double Mini PET With Standard vs. Adapted Dwell Volume and Dwell Time - Proof of Concept of Adapted PD
Brief Title: Proof of Concept of Adapted PD in Children (PC-AAPD)
Acronym: PC-AAPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Hôpital de Hautepierre (Other)
Responsible Party: Principal Investigator, Claus Peter Schmitt, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: S-545/2015
Record Dates: First submitted 2016-04-13; First posted 2016-04-22 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Primary Study Outcome: Sodium Clearance in Dialysis; Solute Removal; Ultrafiltration
Keywords: Adapted APD; Dialytic Sodium Removal; Ultrafiltration; Clearance rate; Intraperitoneal pressure
MeSH Terms: interventions — Peritoneal Dialysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapted double mini PET (Active Comparator): PET = Peritoneal Equilibration Test, a test routinely performed to measure peritoneal transport rates of solutes and water in peritoneal dialysis patients. To this end the routinely administered dialysis fluid is infused into the peritoneal cavity. The test will be modified (adapted):
  A short, small cycle (0.6 mL/m² BSA, 30 min) followed by a long, large cycle (1.4 mL/m², 120 min) will be performed in each patient and compared to a standard double mini PET.
  Interventions: Other: Adapted double mini PET
- Standard double mini PET (Placebo Comparator): The Standard double mini PET consists of two identical cycles (fill volume 1 L/m², 75 min of dwell time)
  Interventions: Other: Standard double mini PET

INTERVENTIONS:
Other: Adapted double mini PET — The modified double mini PET mimics the treatment of adapted PD and thus allows its validation
  Other Names: Peritoneal Equilibration Test (PET); Peritoneal dialysis
  Arms: Adapted double mini PET
Other: Standard double mini PET — The standard double mini PET reflects the routine PD treatment in children and is used for standardized comparison
  Other Names: Peritoneal Equilibration Test (PET); Peritoneal dialysis
  Arms: Standard double mini PET

SUMMARY:
The purpose of this study is to validate the concept of adapted automated PD a modified Peritoneal Equilibration Test (PET), will be performed in children on chronic PD. Instead of a single 4 hour standard dwell, two double mini PET using the same type and total volume of dialysate and the same total dwell time (150min) will be performed in randomised sequence. An double mini test consists of two identical dwells, reflecting routine PD, the other one of a short small dwell followed by a long, large dwell as suggested from adapted PD regimes successfully applied in adult PD patients.

DETAILED DESCRIPTION:
Present peritoneal dialysis treatment is hampered by the limited efficacy of currently applied regimen, mainly consisting of a series of standard dwells with the same amount of dialysate and dwell time. New cycler machines available for routine therapy now allow modification of time and volume of each dwell and thus to individually adapt PD regime. In fact a recent multi-center trial in adult patients suggests that a PD regimen consisting of a sequence of short small dwells followed by large and long lasting dwells in total applying the same amount of dialysate during the same total treatment time substantially improves fluid and toxin removal. Underlying beneficial mechanisms are highly debated. Prior to adaptation of such PD treatment patterns to children on automated PD in the routine clinical setting, the tolerability and biochemical effects need to be demonstrated.

To this end, the Peritoneal Equilibration Test (PET), which is routinely performed in children during a day hospital treatment to analyse peritoneal transport function, will be modified. Instead of a single 4 hour standard dwell, two double mini PET using the same type and total volume of dialysate and the same total dwell time (150min) will be performed in randomised sequence in a total of 15 stable pediatric PD patients treated in four different European pediatric dialysis centres. The conventional double mini PET consists of two identical cycles (fill volume 1 L/m², 75 min), the adapted one of a short, small cycle (0.6 mL/m² BSA, 30 min) followed by a long, large cycle (1.4 mL/m², 120 min). A total of 22 ml of blood will be drawn via a peripheral i.v. line, intraperitoneal pressure, in clinical routine controlled once during a PET, will be measured with each dwell.

The study analyses the time and volume dependent PD transport mechanisms. Patients included may benefit from the detailed analysis of peritoneal membrane function, allowing for optimisation of the individual PD prescription.

ELIGIBILITY:
Inclusion Criteria:

* PD patients 5-21 years of age
* Stable PD
* Last peritonitis > 4 weeks ago

Exclusion Criteria:

* Polyuria and dehydrated patients (as to the clinical status RR, HR and BCM) not allowing for more than 1.5% glucose content of PD fluid
* Hypoalbuminemia (serum albumin < 25g/l)
* Relevant changes in dialysis regime and diet the three days preceding the study
* Hb < 9 mg/dl
* Pregnancy
* History of repeated hernia or PD fluid leakage
* Intolerability of intraperitoneal pressure of up to 18 cm H2O at 1400ml/m²
* BSA in supine position (e.g. due to organomegaly)
* Any underlying diseases affecting the peritoneal membrane transport function (such as previous surgery with subsequent adhesions and fluid trapping, chronic bowl disease)
* Heart insufficiency
* Patients with catheter dysfunction, i.e. outflow problems (assessed by cycler alarms during the last 2 weeks)

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Dialytic sodium removal, i.e. the amount of sodium (mmol) per double mini PET (via ultrafiltration and diffusive sodium transport) | 2 x 150 min with one 1 hour inbetween each PET
  two double mini PET each comprising 150 min of dialysis

SECONDARY OUTCOMES:
dialytic water and solute removal, i.e. ultrafiltrate per double mini PET (ml/gram intraperitoneal glucose exposure), phosphate removal per dmPET (mmol); Kt/V, clearance of creatinine (ml/min*1.73m²), intraperitoneal pressure (cm water) | 2 x 150 min with one 1 hour inbetween each PET
  two double mini PET each comprising 150 min of dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Claus P Schmitt, MD, Principal Investigator — Center for Pediatric and Adolescent Medicine
Locations (1):
- Center for Pediatric and Adolescent Medicine, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fischbach M, Schmitt CP, Shroff R, Zaloszyc A, Warady BA. Increasing sodium removal on peritoneal dialysis: applying dialysis mechanics to the peritoneal dialysis prescription. Kidney Int. 2016 Apr;89(4):761-6. doi: 10.1016/j.kint.2015.12.032. Epub 2016 Jan 21. PMID 26924063
- [Result] Fischbach M, Zaloszyc A, Schaefer B, Schmitt CP. Optimizing peritoneal dialysis prescription for volume control: the importance of varying dwell time and dwell volume. Pediatr Nephrol. 2014 Aug;29(8):1321-7. doi: 10.1007/s00467-013-2573-x. Epub 2013 Aug 2. PMID 23903692
- [Result] Fischbach M, Issad B, Dubois V, Taamma R. The beneficial influence on the effectiveness of automated peritoneal dialysis of varying the dwell time (short/long) and fill volume (small/large): a randomized controlled trial. Perit Dial Int. 2011 Jul-Aug;31(4):450-8. doi: 10.3747/pdi.2010.00146. Epub 2011 Mar 31. PMID 21454393